CLINICAL TRIAL: NCT02083783
Title: TRI102 in the Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHA): A Laboratory Classroom Study
Brief Title: TRI102 in the Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRI102-ADD-001
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — TRI102 protein, Gibberella zeae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRI102 (Experimental): Active, amphetamine extended-release oral suspension
  Interventions: Drug: TRI102
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TRI102 — formulation containing active moiety (amphetamine)
  Other Names: amphetamine extended-release oral suspension
  Arms: TRI102
Other: Placebo — formulation without active moiety
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether TRI102 is effective in the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in children ages 6-12.

DETAILED DESCRIPTION:
A Phase 3, randomized, double-blind, placebo-controlled, parallel group, multicenter, laboratory classroom study. After Screening and Baseline evaluations, eligible subjects are enrolled in the study and entered the open-label phase, dose-optimization phase. TRI102 is taken once daily and subjects undergo dose optimization activities for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years with ADHD who require pharmacologic treatment for this condition

Exclusion Criteria:

* Other serious illnesses or conditions that would put the patient at particular risk for safety events or would interfere with treatment/assessment of ADHD

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wigal, PhD, Principal Investigator — Newport Beach Clinical Research Associates, Inc.
Locations (5):
- United States (5):
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Bayou City Research, Houston, Texas
  - Westex Clinical Investigation, Lubbock, Texas

REFERENCES:
- [Derived] Faraone SV, Childress AC, Gomeni R, Rafla E, Kando JC, Dansie L, Naik P, Pardo A. Efficacy of Amphetamine Extended-Release Oral Suspension in Children with Attention-Deficit/Hyperactivity Disorder: Effect Size Across the Day. J Child Adolesc Psychopharmacol. 2023 Feb;33(1):14-19. doi: 10.1089/cap.2022.0093. Epub 2023 Feb 2. PMID 36730749

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 subjects not randomized.
Groups:
- TRI102: Active
  TRI102: formulation containing active moiety
  The stable dose of TRI102 reached during the Dose Optimization Period varied between 10 to 20 mg/day and was determined based on Investigator clinical judgment and assessments of both tolerability and efficacy for each subject. The same stable dose identified for a subject during the Dose Optimization Period was administered during the double-blind Treatment Period.
- Placebo: Placebo
  Placebo: formulation without active moiety
  The same stable dose identified for a subject during the Dose Optimization Period was administered during the double-blind Treatment Period.
Period: Overall Study
Arm/Group | TRI102 | Placebo
Started (Open-Label Optimization) | 52 | 48
Completed | 51 | 48
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | TRI102 | Placebo | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.2 (1.95) | 9.6 (1.76) | 9.4 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 36 | 32 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 33 | 27 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 15 | 34
  White | 27 | 28 | 55
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
ADHD Type [Count of Participants; unit: Participants]
  Predominantly inattentive | 12 | 8 | 20
  Predominantly impulsive | 0 | 1 | 1
  Combined | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: SKAMP (Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale)
Description: Change from baseline in SKAMP-Combined Scores measured approximately 4 hours after dose (active or placebo). The SKAMP-Combined score is obtained by summing 13 assessment items, where each item is rated on a 7-point scale (0 = normal to 6 = maximal impairment). This gives an overall (combined) SKAMP Score of 0= normal to 78 which indicates maximal impairment. The endpoint is assessed as a change from baseline in the overall score on the 78-point scale.
Time Frame: Absolute change from baseline in SKAMP-C score from baseline to 4 hours after dose
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TRI102 | Placebo
Number analyzed (Participants) | 51 | 48
score on a scale | -9.1 (7.51) | 5.6 (7.85)
Statistical Analysis 1: Comparison: TRI102 vs Placebo; Treatment difference in SKAMP-C scores from baseline to 4 hours postdose; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.68, 95% CI 2-sided [-17.9 to 11.6]

2. Secondary Outcome: PERMP (Permanent Product Measure of Performance).
Description: The PERMP is a math test that measures effortful performance without a learning curve (Wigal and Wigal 2006). The test determines the number of problems attempted and the number of problems correctly answered. In this study, the primary efficacy measure was a PERMP evaluation done 4 hours after taking study medication, a time selected a priori to coincide with the known pharmacodynamic effects based on prior research and to minimize the impact of repeated measures on adjustment of multiplicity (Wigal et al. 1998; Pelham et al. 2001). The PERMP consists of 400 math questions and each are scored. PERMP scores are expressed as the number of questions correct. Predose PERMP Tests are compared with post-dose PERMP scores at prespecfied timepoints.
Time Frame: Absolute change from baseline in PERMP questions answered correctly, measured from baseline to 4 hours postdose.
Population: Intention to treat
Measure: Least Squares Mean (Standard Error); unit: PERMP questions answered correctly
Arm/Group | TRI102 | Placebo
Number analyzed (Participants) | 51 | 48
PERMP questions answered correctly | 25.3 (4.21) | -13.6 (4.39)
Statistical Analysis 1: Comparison: TRI102 vs Placebo; p-value for comparison between change from baseline in placebo vs active treatment; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 38.9, 95% CI 2-sided [27.3 to 50.6]

ADVERSE EVENTS:
Time Frame: Screening through Follow up (9 weeks)
Description: AEs were recorded at each study visit for a total of 9 weeks.
Arm/Group | TRI102 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 6/52 | 1/48
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRI102 (N=52) | Placebo (N=48)
Abdominal pain, upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis, allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No